CLINICAL TRIAL: NCT03378258
Title: Petechiae In Children (PIC) Study
Brief Title: Petechiae In Children (PIC) Study: Defining A Clinical Decision Rule for The Management Of Fever and Non-Blanching Rashes In Children Including The Role Of Point Of Care Testing For Procalcitonin & Neisseria Meningitidis DNA.
Acronym: PIC
Status: Completed | Type: Observational
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Pediatric Emergency Research in the UK and Ireland (PERUKI) (Other); Royal College of Emergency Medicine (Other); Queen's University, Belfast (Other); Public Health Agency (Northern Ireland) (Unknown)
Responsible Party: Sponsor
Other Study IDs: EAT/5313/16; 17/NI/0169 (Other: Research Ethics Committee)
Record Dates: First submitted 2017-11-27; First posted 2017-12-19 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Meningitis, Meningococcal; Meningococcal Sepsis; Meningococcal Disease; Meningococcal Infections; Sepsis; Meningitis
Keywords: meningococcal; neisseria meningitidis; sepsis; meningitis; procalcitonin; PCT; LAMP; loop-mediated-isothermal AMPlification
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections; Sepsis; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma for testing of biomarkers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A fever and a non-blanching rash is a relatively common reason for a child to attend an emergency department. A fever and a non-blanching rash can be an early sign of a life-threatening infection known as meningococcal disease. The aim of the PIC study is to determine how best to diagnose early meningococcal disease in children.

In particular the investigators are interested in researching how quick bedside tests can be used to do this.

DETAILED DESCRIPTION:
A fever an a non-blanching rash is a relatively common presentation the the emergency department. A minority of children with a fever and a non-blanching rash with have a life-threatening infection. Currently it is very difficult to determine those children that require urgent treatment from those that have a simple viral illness.

The aim of the PIC study is to research how to better diagnose those serious infections earlier.

Data from the study will be used to test the effectiveness of current practice and to identify areas where current practice could be improved.

ELIGIBILITY:
Inclusion Criteria:

* Fever (recorded or reported) 38 degrees Centigrade or higher and a non-blanching rash (at the time of presentation)
* Features of meningococcal sepsis/meningitis

Exclusion Criteria:

* Known haematological conditions such as haematological malignancy, idiopathic thrombocytopenic purpura and coagulopathy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All Children <18 years of age (male and female) attending with a fever (recorded or reported) 38C and a non-blanching rash (at the time of presentation) or features of meningococcal sepsis/meningitis will be eligible for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 1329 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Confirmation of meningococcal infection | 72 hours from testing
  Blood and Cerebrospinal fluid (CSF) culture or quantitative Polymerase Chain Reaction (PCR) will be used to confirm meningococcal infection

CONTACTS AND LOCATIONS:
Overall Officials: MIchael D Shields, Principal Investigator — Queen's University, Belfast
Locations (1):
- Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data requests will be reviewed by an external independent review panel. Requesters will be required to sign a data access agreement.

REFERENCES:
- [Background] Meningitis Research Foundation. Meningococcal Meningitis and Septicaemia. 2016. https://www.meningitis.org/getmedia/cf777153-9427-4464-89e2-fb58199174b6/gp_booklet-UK-sept-16. Accessed 10 Oct 2017.
- [Background] O Maoldomhnaigh C, Drew RJ, Gavin P, Cafferkey M, Butler KM. Invasive meningococcal disease in children in Ireland, 2001-2011. Arch Dis Child. 2016 Dec;101(12):1125-1129. doi: 10.1136/archdischild-2015-310215. Epub 2016 Aug 26. PMID 27566800
- [Background] Meningitis (bacterial) and meningococcal septicaemia in under 16s: recognition, diagnosis and management. London: National Institute for Health and Care Excellence (NICE); 2015 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK555182/ PMID 32207890
- [Background] Bourke TW, McKenna JP, Coyle PV, Shields MD, Fairley DJ. Diagnostic accuracy of loop-mediated isothermal amplification as a near-patient test for meningococcal disease in children: an observational cohort study. Lancet Infect Dis. 2015 May;15(5):552-8. doi: 10.1016/S1473-3099(15)70038-1. Epub 2015 Feb 27. PMID 25728843
- [Background] Brogan PA, Raffles A. The management of fever and petechiae: making sense of rash decisions. Arch Dis Child. 2000 Dec;83(6):506-7. doi: 10.1136/adc.83.6.506. PMID 11087287
- [Background] Mandl KD, Stack AM, Fleisher GR. Incidence of bacteremia in infants and children with fever and petechiae. J Pediatr. 1997 Sep;131(3):398-404. doi: 10.1016/s0022-3476(97)80065-0. PMID 9329416
- [Background] Nielsen HE, Andersen EA, Andersen J, Bottiger B, Christiansen KM, Daugbjerg P, Larsen SO, Lind I, Nir M, Olofsson K. Diagnostic assessment of haemorrhagic rash and fever. Arch Dis Child. 2001 Aug;85(2):160-5. doi: 10.1136/adc.85.2.160. PMID 11466193
- [Background] Riordan FA, Jones L, Clark J; Non-Blanching Rash Audit Group. Validation of two algorithms for managing children with a non-blanching rash. Arch Dis Child. 2016 Aug;101(8):709-13. doi: 10.1136/archdischild-2015-309451. Epub 2016 Mar 16. PMID 26984401
- [Derived] Waterfield T, Maney JA, Fairley D, Lyttle MD, McKenna JP, Roland D, Corr M, McFetridge L, Mitchell H, Woolfall K, Lynn F, Patenall B, Shields MD; Paediatric Emergency Research in the UK and Ireland (PERUKI) Group. Validating clinical practice guidelines for the management of children with non-blanching rashes in the UK (PiC): a prospective, multicentre cohort study. Lancet Infect Dis. 2021 Apr;21(4):569-577. doi: 10.1016/S1473-3099(20)30474-6. Epub 2020 Nov 10. PMID 33186517
- [Derived] Waterfield T, Maney JA, Lyttle MD, McKenna JP, Roland D, Corr M, Patenall B, Shields MD, Woolfall K, Fairley D; Paediatric Emergency Research in the UK and Ireland (PERUKI). Diagnostic test accuracy of point-of-care procalcitonin to diagnose serious bacterial infections in children. BMC Pediatr. 2020 Oct 21;20(1):487. doi: 10.1186/s12887-020-02385-2. PMID 33087092
- [Derived] Waterfield T, Lyttle MD, McKenna J, Maney JA, Roland D, Corr M, Woolfall K, Patenall B, Shields M, Fairley D; Paediatric Emergency Research in the UK and Ireland (PERUKI). Loop-mediated isothermal amplification for the early diagnosis of invasive meningococcal disease in children. Arch Dis Child. 2020 Dec;105(12):1151-1156. doi: 10.1136/archdischild-2020-319139. Epub 2020 Jun 25. PMID 32586928
- [Derived] Waterfield T, Lyttle MD, Shields M, Fairley D, Roland D, McKenna J, Woolfall K; Paediatric Emergency Research in the UK and Ireland (PERUKI). Parents' and clinicians' views on conducting paediatric diagnostic test accuracy studies without prior informed consent: qualitative insight from the Petechiae in Children study (PiC). Arch Dis Child. 2019 Oct;104(10):979-983. doi: 10.1136/archdischild-2019-317117. Epub 2019 Jun 7. PMID 31175126
- [Derived] Waterfield T, Lyttle MD, Fairley D, Mckenna J, Woolfall K, Lynn F, Maney JA, Roland D, Weir A, Shields MD; Paediatric Emergency Research in the UK and Ireland (PERUKI). The "Petechiae in children" (PiC) study: evaluating potential clinical decision rules for the management of feverish children with non-blanching rashes, including the role of point of care testing for Procalcitonin & Neisseria meningitidis DNA - a study protocol. BMC Pediatr. 2018 Jul 30;18(1):246. doi: 10.1186/s12887-018-1220-x. PMID 30060751